CLINICAL TRIAL: NCT01624922
Title: The China PEACE (Patient-centered Evaluative Assessment of Cardiac Events) Prospective Study of Percutaneous Coronary Intervention
Brief Title: China PEACE-Prospective PCI Study
Status: Completed | Type: Observational
Sponsor: China National Center for Cardiovascular Diseases (Other Government)
Collaborators: Ministry of Health, China (Other Government)
Responsible Party: Sponsor
Other Study IDs: WSGY-201202025-4
Record Dates: First submitted 2012-06-17; First posted 2012-06-21 (Estimated); Last update posted 2015-08-31 (Estimated); Status verified 2015-08

CONDITIONS: Coronary Heart Disease
MeSH Terms: conditions — Coronary Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — A venous blood sample of 20mL will be collected at 1-month visit and 12-month visit for biomarker analysis and storage for future genetic studies;
  A urine samples of 40mL will be collected at 1-month visit and 12-month visit for biomarker analysis and storage.
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Coronary heart disease (CHD) pose a serious health threaten to population. PCI, as a well-proved and booming measure in CHD management, is invasive and of high cost, however the knowledge about the real-life PCI use in China is limited. By consecutively recruiting PCI patients in 30 geographically representative highest-rank hospitals, this study will examine various real-life factors, that may affect patients recovery after the procedure. Practical guidelines, appropriateness criteria and quality evaluative system for PCI will be established based on the findings, to improve patients outcomes in future finally.

DETAILED DESCRIPTION:
Cardiovascular disease (CVD) is a major concern in public health globally, as well as in China, and remarkable variations of resources available and health system performance have been noted. Relatively limited information is available about how evidence-based therapies are incorporated appropriately into routine clinical practice. In addition, little information is available about the magnitude and quality of PCI, which has developed rapidly during the past several decades. Practical and applied knowledge from large unselected population is needed to guide practice and policy for quality improvement and cost reduction.

This study will enroll patients undergoing PCI after admission consecutively in 30 tertiary hospitals scattered all over China. At study entry, participants will be interviewed during their index hospitalization, to collect information about symptoms, functioning, quality of life, and medical care. Demographic characteristics, medical history, clinical features, diagnostic tests, medications, procedures, and in-hospital outcomes of patients will be abstracted from medical records by well trained professional abstractors. And CAG imaging will be reviewed by national and international expert panels. At 1 month, 6 month, and 12 month after discharge, participants will return to the clinic for follow up visits, a face-to-face interview will be conducted to get information about clinical events, symptoms, functioning, quality of life, and medical care during the recovery period. At 1-Month and 12-Month follow-up visit, blood and urine sample will be collected. Participants' blood samples will be stored for future biologic and genetic studies. This study will examine various real-life factors that may affect patients recovery after PCI, including patients' characteristics and treatment measures. Practical guidelines, quality evaluative system, and appropriateness criteria will be established based on the findings, to improve patients outcomes in future finally.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized patients undergoing a percutaneous coronary intervention (PCI) with stents implantation for coronary lesions.

Exclusion Criteria:

* Previously enrolled in the PEACE study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: In 30 tertiary hospitals with capability of Percutaneous Coronary Intervention in China, 3000 hospitalized patients undergoing Percutaneous Coronary Intervention will be enrolled consecutively.
Sampling Method: Non-Probability Sample
Enrollment: 5185 (Actual)
Dates: Start 2012-12; Primary Completion 2013-08 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Major adverse cardiovascular events (MACE) | 1 year
  Composite of major adverse cardiovascular events (MACE) including cardiac death, non-fatal AMI, coronary revascularization procedure, or ischemic stroke.

SECONDARY OUTCOMES:
Symptoms status (SAQ) | 1 year
Quality of life (EQ-5D) | 1 year
Depression (PHQ-8) | 1 year
Stress (PSS-4) | 1 year
Cardiac death | 1 year
Fatal or non-fatal AMI | 1 year
Coronary revascularization procedure | 1 year
Ischemic stroke | 1 year
Re-admission | 1 year
Adherence to medications for secondary prevention | 1 year
  Taking the following medications for 6 or more days per week: aspirin, clopidogrel, ACEI/ARB, statin and beta-blockers
Control of risk factors | 1 year
  Control of hypertension, diabetes, dyslipidemia, smoking, and obesity

OTHER OUTCOMES:
Cognitive function (MMSE) | 1 year
Sexual activity/function | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Lixin Jiang, M.D., Ph.D., Principal Investigator — China National Center for Cardiovascular Diseases; Harlan M Krumholz, M.D., S.M., Principal Investigator — Yale University
Locations (1):
- Fuwai Hospital, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Zheng X, Dreyer RP, Curtis JP, Liu S, Xu X, Bai X, Li X, Zhang H, Wang S, Masoudi FA, Spertus JA, Li J, Krumholz HM; China PEACE Collaborative Group. Sex Differences in 1-Year Health Status Following Percutaneous Coronary Intervention in Patients Without Acute Myocardial Infarction: Results From the China PEACE Prospective Study. J Am Heart Assoc. 2020 Mar 17;9(6):e014421. doi: 10.1161/JAHA.119.014421. Epub 2020 Mar 5. PMID 32131687